CLINICAL TRIAL: NCT06962215
Title: The Impact of Paramedic Training in Simulation on the Experience of Patients Treated for Malignant Brain Tumors in Neurosurgery
Brief Title: The Impact of Paramedic Training in Simulation on the Experience of Patients Treated for Malignant Brain Tumors in Neurosurgery (IPSIMANON)
Acronym: IPSIMANON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 29BRC24.0039 - IPSIMANON; 2024-A00353-44 (Other: Agence Nationale de Sécurité du Médicament et des produits de santé (ID-RCB))
Record Dates: First submitted 2025-03-26; First posted 2025-05-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Brain Tumor Adult
Keywords: Brain tumor; Simulation Training; Paramedical; Neurosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Cluster randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Centers whose paramedics will not follow the training proposed by the study.
- Paramedic training (Experimental): Centers whose paramedics will benefit from the training proposed by the study.
  Interventions: Other: Paramedic training

INTERVENTIONS:
Other: Paramedic training — Nurses and care assistants at the centers randomized to the "with training" arm will undergo a day-and-a-half of training to help them support patients diagnosed with brain tumors. Training consists of half a day of theory, followed by a day of simulation.
  Arms: Paramedic training

SUMMARY:
The goal of this clinical trial is to demonstrate that simulation training for paramedical staff in neurosurgery departments, in announcing and accompanying patients with a brain tumor, improves patient satisfaction when a (potentially malignant) brain tumor is discovered, compared with usual care.

The main question it aims to answer is:

- Are patients more satisfied (as measured by scores on the EORCT IN-PATSAT32 questionnaire) with their neurosurgical hospitalization following the discovery of a brain tumor in centers where paramedics have been trained by simulation?

Researchers will compare the results of the EORTC IN-PATSAT32 questionnaire to determine whether paramedic training improves patient satisfaction between simulation-trained and untrained centers.

Participants will be asked to complete the EORT IN-PATSAT32 questionnaire at the end of their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient covered by a social security scheme
* Patient signed informed consent form
* Patient found to have a brain tumor (potentially malignant, primary or secondary if this is the mode of entry into the disease)
* Hospitalization in the Neurosurgery Department at the time of tumor discovery, before the histological diagnosis is announced.

Exclusion Criteria:

* Patients with a personal history of cancer
* Patient without family AND unable to receive information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Measuring patient satisfaction following the discovery of a brain tumor. | The day of discharge from neurosurgery, on average 8 days (between 1 days and 15 days)
  Measurement of patient satisfaction following the discovery of a brain tumor via scores obtained, at the end of their neurosurgical hospitalization, in response to the EORCT IN-PATSAT32 (European Organisation of Research and Treatment of Cancer IN PATient SATisfaction 32) questionnaire, whose dimensions of interest are ordered as follows for hierarchical analysis:
  1. SATNIS = nurses interpersonal skills
  2. SATNIP = nurses information provision
  3. SATNAV = nurses availability
  4. SATNTS = nurses technical skills,
  5. SATGEN = overall quality rating All of the scales and single-item measures range in score from 0 to 100. A high score represents a high level of satisfaction with care.

SECONDARY OUTCOMES:
Measurement of patients' experiences following the discovery of a brain tumor via scores obtained (other questionnaire items) | The day of discharge from neurosurgery, on average 8 days (between 1 days and 15 days)
  Measurement of patients' experiences following the discovery of a brain tumor via the scores obtained at the end of their neurosurgical hospitalization in response to the other items of the EORTC IN-PATSAT32 questionnaire (European Organisation of Research and Treatment of Cancer IN PATient SATisfaction 32) :
  * SATEXE = exchange of information between caregivers,
  * SATDIS = doctors interpersonal skills,
  * SATDIP = doctors information provision,
  * SATDAV = doctors availability,
  * SATDTS = doctors technical skills,
  * SATOTH = other personal interpersonal skills, All of the scales and single-item measures range in score from 0 to 100. A high score represents a high level of satisfaction with care.
Measuring patients' feelings | The day of discharge from neurosurgery, on average 8 days (between 1 days and 15 days)
  Measuring patients' feelings with the INCA (French National Cancer Institute) questionnaire (Sick people - Survey on the announcement of the diagnosis and the feelings of sick people) at the end of their neurosurgical hospital hospitalization.
Measuring Caregivers' Experiences/Quality of Life at Work | Day 0 and Month 6
  Measurement of caregivers' experience/quality of life at work at D0 and 6 months, using the Delmas et al. questionnaire.
Measurement of caregivers' listening skills. | Day 0, after training and Month 6
  Measurement of caregivers' listening attitude, using the Porter et al. questionnaire at D0, after training and 6 months.
Measuring communication within the paramedical team | Day 0 and Month 6
  Measurement of communication within the paramedical team, using the paramedical team communication evaluation questionnaire (Likert scales, 5 points) at D0 and 6 months.
Measuring communication between paramedical and medical teams. | Day 0 and Month 6
  Measurement of communication between the paramedical and medical teams, using a questionnaire to evaluate communication between the paramedical and medical teams (Likert scales, 5 points) at D0 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie QUEMENEUR, Study Director — CHU Brest
Locations (11):
- France (11):
  - CHU Brest, Brest, Brittany Region
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - APHM Nord, Marseille
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available from five years to fifteen years after completion of the final study report.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.